CLINICAL TRIAL: NCT06554028
Title: Tislelizumab and Induction Chemotherapy Followed by Radiotherapy or Adaptive Surgery for Larynx Preservation in Resectable Locally Advanced Laryngeal or Hypopharyngeal Cancer: A Single-Arm Phase II Clinical Trial
Brief Title: Tislelizumab and Induction Chemotherapy for Larynx Preservation in Resectable Advanced Laryngeal/Hypopharyngeal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-192
Record Dates: First submitted 2024-08-05; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-07

CONDITIONS: Laryngeal Cancer; Hypopharynx Cancer; Laryngeal Neoplasms
MeSH Terms: conditions — Laryngeal Neoplasms; Hypopharyngeal Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tislelizumab and Induction Chemotherapy Followed by Radiotherapy or Adaptive Surgery (Experimental): Induction chemotherapy TP regimen combined with Tislelizumab for 3 cycles: Cisplatin 37.5mg/m2 d1-2 q3w, Docetaxel 37.5mg/m2 d1and d3 q3w,Tislelizumab 200mg d3 q3w.
  Response rate of primary tumor or lymph nodes is evaluated using laryngoscopy and head and neck MRI after 3 cycles of induction therapy. If the primary lesion reaches CR/PR and the lymph nodes reach CR, chemoradiotherapy based on cisplatin is conducted. If the primary lesion reaches CR/PR and lymph node PR/PD, cervical lymph node dissection will be performed, followed by radiotherapy/concurrent chemoradiotherapy. If the primary lesion is SD/PD, regardless of the condition of the lymph nodes, primary lesion resection and lymph node dissection should be performed, followed by adjuvant radiation/chemoradiation.
  Interventions:
  Drug: chemotherapy TP regimen combined with Tislelizumab
  Interventions: Drug: chemotherapy TP regimen combined with Tislelizumab

INTERVENTIONS:
Drug: chemotherapy TP regimen combined with Tislelizumab — Induction chemotherapy TP regimen combined with Tislelizumab for 3 cycles: Cisplatin 37.5mg/m2 d1-2 q3w, Docetaxel 37.5mg/m2 d1and d3 q3w,Tislelizumab 200mg d3 q3w.
  •Response rate of primary tumor or lymph nodes is evaluated using laryngoscopy and head and neck MRI after 3 cycles of induction therapy. If the primary lesion reaches CR/PR and the lymph nodes reach CR, chemoradiotherapy based on cisplatin is conducted. If the primary lesion reaches CR/PR and lymph node PR/PD, cervical lymph node dissection will be performed, followed by radiotherapy/concurrent chemoradiotherapy. If the primary lesion is SD/PD, regardless of the condition of the lymph nodes, primary lesion resection and lymph node dissection should be performed, followed by adjuvant radiation/chemoradiation.
  Other Names:
  Docetaxel Cisplatin Paclitaxel

SUMMARY:
This study is a prospective, single-arm, single-center, phase II study. The goal of this clinical trial is to explore the therapeutic value of the treatment model of "tislelizumab combined with chemotherapy followed by radiotherapy/adaptive surgery" on larynx Preservation of locally advanced hypopharyngeal cancer and laryngeal cancer.

DETAILED DESCRIPTION:
Historical studies have shown that induction chemotherapy can provide an opportunity to preserve the larynx in approximately 60-70% of patients with locally advanced laryngeal/hypopharynx carcinoma. Recently, phase I-II clinical studies have shown that induction of PD-1 inhibitors has a good pathological response in locally advanced head and neck cancer, with or without combined chemotherapy. However,the primary lesion and lymph nodes respond asynchronously or even in the opposite way to immune induction therapy. The primary lesion is more likely to achieve CR/PR, while the lymph nodes are more likely to show PR/SD or even PD. Therefore, the surgical or radiotherapy plan should be implemented according to the specific response of the primary lesion and metastatic lymph nodes to induction therapy. This study aimed to determine whether the combination of induction chemotherapy with a PD-1 inhibitor (Tislelizumab) followed by chemoradiotherapy or adaptive surgery can improve the rate of laryngeal preservation in patients with resectable laryngeal/hypopharynx cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed, resectable locally advanced laryngeal/hypopharyngeal squamous cell carcinoma (T2-4a, N0-resectable N3, M0);
2. Age between 18-70 years;
3. Had at least one measurable lesion according to RECIST 1.1 criteria;
4. Anticipated overall survival more than 3 months;
5. Satisfactory performance status: ECOG (Eastern Cooperative Oncology Group) scale 0-1;
6. Normal organ function;
7. Male and no pregnant female, able to adapt birth control methods during treatment;
8. Signed inform consent;

Exclusion Criteria:

1. Hypersensitivity to tislelizumab, Paclitaxel or Cisplatin.
2. Received anti-tumor treatment in the past 6 months, including radiotherapy and chemotherapy, surgery, immunotherapy.
3. Suffered from malignant tumors, except cervical carcinoma in situ, papillary thyroid carcinoma, or skin cancer (non- melanoma) within five years.
4. There is distant metastasis.
5. Active autoimmune diseases, history of autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); but excludes autoimmune-mediated hypothyroidism on stable doses of thyroid replacement hormone; type 1 diabetes on stable doses of insulin; vitiligo or resolved childhood asthma/allergies, Patients who do not require any intervention after adulthood.
6. Known history of primary immunodeficiency (including positive HIV test, or suffering from other acquired or congenital immunodeficiency diseases, or history of organ transplantation and allogeneic bone marrow transplantation);
7. Severe infection occurred within 4 weeks before the first use of the study drug, such as severe pneumonia requiring hospitalization, bacteremia, infection complications, etc.
8. The subject has severe liver and kidney dysfunction, HIV infection, HCV infection, uncontrolled clinical symptoms or diseases of the heart, such as: heart failure above NYHA grade II or echocardiography，showing left ventricular ejection fraction (LVEF) < 50%; unstable angina; myocardial infarction within 1 year; patients with clinically significant supraventricular or ventricular arrhythmias requiring clinical，intervention (including QTc interval ≥ 470 ms); uncontrolled diabetes, uncontrolled Patients with high blood pressure, hypertensive crisis or hypertensive encephalopathy or other diseases considered by the researchers to be ineligible.
9. Patients with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) DNA exceeding 500 IU/ml, or patients with active hepatitis C virus (HCV) should be excluded; inactive hepatitis B surface Antigen carriers, treated and stable hepatitis B patients (HBV DNA<500IU/ml), and cured hepatitis C patients can be enrolled.
10. Have a history of interstitial lung disease (excluding radiation pneumonitis that has not been treated with hormones) and non-infectious pneumonia.
11. Active tuberculosis infection was found through medical history or CT examination, or patients with a history of active tuberculosis infection within 1 year before enrollment, or patients with a history of active tuberculosis infection more than 1 year ago but without formal treatment.
12. Patients who have received any of the following treatments (1) Subjects who need to be given corticosteroids (> 10 mg prednisone equivalent dose per day) or other immunosuppressants for systemic treatment within 2 weeks before the first use of the study drug, except for local inflammation and prevention of allergies and nausea, Cases of use of corticosteroids for vomiting. In the absence of active autoimmune disease, corticosteroid replacement with inhaled or topical steroids and curative doses of prednisone >10 mg/day is permitted; (2) Have been vaccinated against tumors; those who have been vaccinated or have been vaccinated with live vaccines within 4 weeks before the first administration of the study drug; (3) Received major surgery or severe trauma within 4 weeks before the first use of the study drug; (4) Enrolled in another clinical study at the same time.
13. Pregnant and lactating women. Women of childbearing age must take a pregnancy test within 7 days before enrollment Negative.
14. Substance abuse, clinical or psychological or social factors that hinder informed consent or research conduct influences.
15. Any uncertain factors affecting the safety or compliance of the subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Laryngeal preservation rate at 3 months after radiotherapy | 3-month post-radiotherapy
  defined as the absence of any residual disease that would justify salvage total laryngectomy

SECONDARY OUTCOMES:
Objective response rate after induction chemoimmunotherapy | 2 weeks after the end of cycle 3 of induction therapy
  2 weeks after the 3th cycle of induction therapy
Overall survival rate at 1 year | One year post-radiotherapy
  Overall survival rate at 1 year
Laryngeal preservation rate at 1 year after radiotherapy | 1 year post-radiotherapy
  defined as the absence of any residual disease that would justify salvage total laryngectomy
Progression-free survival rate at 1 year | One year post-radiotherapy
  Progression-free survival rate at 1 year
Pathological complete response rate of the patients receiving surgical resection | Within 3 weeks after surgery
  Pathological complete response rate of the patients receiving surgical resection, evaluated by experienced pathologists
Overall survival rate at 2 year | Two year post-radiotherapy
  Overall survival rate at 2 year
Progression-free survival rate at 2 year | Two year post-radiotherapy
  Progression-free survival rate at 2 year
Laryngeal Preservation rate at 2 year | Laryngeal Preservation rate at 2 year
  Two year post-radiotherapy
Adverse Effect | One year post-radiotherapy
  Adverse Effect, evaluated by CTCAE 4.0.03
Major pathologic response rate of the patients receiving surgical resection | Within 3 weeks after surgery
  Major pathologic response rate, defined as no more than 10% of residual viable tumor, evaluated by experienced pathologists

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forastiere AA, Zhang Q, Weber RS, Maor MH, Goepfert H, Pajak TF, Morrison W, Glisson B, Trotti A, Ridge JA, Thorstad W, Wagner H, Ensley JF, Cooper JS. Long-term results of RTOG 91-11: a comparison of three nonsurgical treatment strategies to preserve the larynx in patients with locally advanced larynx cancer. J Clin Oncol. 2013 Mar 1;31(7):845-52. doi: 10.1200/JCO.2012.43.6097. Epub 2012 Nov 26. PMID 23182993
- [Background] Department of Veterans Affairs Laryngeal Cancer Study Group; Wolf GT, Fisher SG, Hong WK, Hillman R, Spaulding M, Laramore GE, Endicott JW, McClatchey K, Henderson WG. Induction chemotherapy plus radiation compared with surgery plus radiation in patients with advanced laryngeal cancer. N Engl J Med. 1991 Jun 13;324(24):1685-90. doi: 10.1056/NEJM199106133242402. PMID 2034244
- [Background] Lefebvre JL, Pointreau Y, Rolland F, Alfonsi M, Baudoux A, Sire C, de Raucourt D, Malard O, Degardin M, Tuchais C, Blot E, Rives M, Reyt E, Tourani JM, Geoffrois L, Peyrade F, Guichard F, Chevalier D, Babin E, Lang P, Janot F, Calais G, Garaud P, Bardet E. Induction chemotherapy followed by either chemoradiotherapy or bioradiotherapy for larynx preservation: the TREMPLIN randomized phase II study. J Clin Oncol. 2013 Mar 1;31(7):853-9. doi: 10.1200/JCO.2012.42.3988. Epub 2013 Jan 22. PMID 23341517